CLINICAL TRIAL: NCT04215341
Title: Feasibility Study for a Multi-centre Trial Investigating Whether Physiotherapy Improves Outcomes for Children With Dysfunctional Breathing
Brief Title: Physiotherapy for Children With Dysfunctional Breathing
Acronym: PhysDB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Children's NHS Foundation Trust (Other)
Collaborators: University of Sheffield (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: SCH/14/011
Record Dates: First submitted 2015-04-23; First posted 2020-01-02 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Dysfunctional Breathing
MeSH Terms: interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): The study contains a single arm. All children participating in the study will receive the primary intervention which is physiotherapy.
  Interventions: Behavioral: Physiotherapy

INTERVENTIONS:
Behavioral: Physiotherapy — A course of breathing retraining delivered by a physiotherapist and practiced by the participant at home.
  Other Names: None - Inhalers and scans are not interventions

SUMMARY:
Dysfunctional breathing in children primarily affects the ability to participate in sport or exercise but can also stop children doing other activities such as playing musical instruments. Clinical experience has shown that physiotherapy (through the use of breathing retraining and other associated techniques) can stop the symptoms of dysfunctional breathing, allowing children to return to normal activities and reduce or stop inhaled medications.

Whilst there is some evidence in adults with this condition to support the use of physiotherapy, there have been no studies carried out in children investigating whether physiotherapy is beneficial for children with dysfunctional breathing.

This study therefore aims to investigate the feasibility of a future large scale multicentre clinical trial designed to investigate whether physiotherapy improves outcomes for children with dysfunctional breathing. The improved management of this common but under recognised condition would lead to significant improvements in the quality of life of children coupled with the reduction in potentially harmful medications.

ELIGIBILITY:
Inclusion Criteria:

Aged 8-16 years Clinical diagnosis of dysfunctional breathing

Exclusion Criteria:

Uncontrolled comorbidities Participant and parents/guardians not fluent in written and spoken English Inability to follow instructions

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 31 (Actual)
Dates: Start 2014-08-04 (Actual); Primary Completion 2016-08-08 (Actual); Study Completion 2016-08-08 (Actual)

PRIMARY OUTCOMES:
Child and parent proxy report versions of the quality of life questionnaire(PedsQL) | 24 months
  To measure participant and parent proxy report of quality of life in the four domains of physical, emotional, social and school functioning

SECONDARY OUTCOMES:
Symptom questionnaire (Nijmegen questionnaire) | 24 months
  To measure the type and frequency of symptoms commonly associated with dysfunctional breathing
Structured light plethysmography (SLP) scan (Thora-3DI) | 24 months
  To objectively measure breathing pattern and rate without influencing these parameters
Reliever inhaler usage recorded using a data logger device | 24 months
  To measure usage of inhaled reliever medication

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Barker, Principal Investigator — Investigator
Locations (1):
- Sheffield Children's NHS Foundation Trust, Sheffield, Sheffield (South Yorkshire District), United Kingdom